CLINICAL TRIAL: NCT04643613
Title: Role of Ready to Drink Nutritional Formula (Protison Enriched With ω-3 FA and BCAA) Supplemented by Nasogastric Tube Feeding in Various Cancer Patients: A Randomized Clinical Trial
Brief Title: Effect of Nutritional Formula (Protison) on Various Cancer Patients: A Randomized Clinical Trial
Acronym: Protison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Chin Kun Wang, Professor, Chung Shan Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS17106
Record Dates: First submitted 2020-11-16; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Cancer
Keywords: Cancer; Cachexia; Nutritional status; Tube feeding; PCNF
MeSH Terms: conditions — Neoplasms; Cachexia

STUDY DESIGN:
Intervention Model Description: Supplementation with the commercial nutritional formula (PCNF; 237 mL/Pack) for 5-6 times/day via bolus NG tube feeding for 12 weeks
Masking Description: None, since treating cancer patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PCNF (Experimental): Totally 42 cancer patients with poor nutritional status under nasogastric (NG) tube feeding was recruited and administered with the commercial nutritional formula (PCNF; 237 mL/Pack) for 5-6 times/day via bolus NG tube feeding for 12 weeks (84 days).
  Interventions: Dietary Supplement: Protison cancer nutritional formula (PCNF)

INTERVENTIONS:
Dietary Supplement: Protison cancer nutritional formula (PCNF) — PCNF (237 mL/Pack) for 5-6 times/day via bolus NG tube feeding for 12 weeks
  Other Names: Protison

SUMMARY:
Many studies (including ASPEN/ESPEN) have demonstrated that balanced diet formula rich in omega 3 fatty acids (ω-3 FA), fibers, protein as well as mineral, vitamins (trace elements) are essential for cancer patients to improve health status and tolerability of chemotherapy. Hence, the present multi-centered, randomized clinical trial was framed to evaluate the efficacy of ready to use balanced nutritional formula-PCNF (rich in ω-3 FA, fibers, MTC, BCAA, and micro-nutrients), in various cancer patient by checking calorie intake and overall health status through assessing various anthropometric and biochemical parameters especially total proteins, pre-albumin, and transferrin.

DETAILED DESCRIPTION:
Many studies (including ASPEN/ESPEN) have demonstrated that balanced diet formula rich in omega 3 fatty acids (ω-3 FA), fibers, protein as well as mineral, vitamins (trace elements) are essential for cancer patients to improve health status and tolerability of chemotherapy. Hence, oncologic nutritionist strongly recommends cancer patients (with cachexia) to consume a diet rich in protein and dietary fibers along with balanced essential micronutrients like vitamins and minerals (Van Norren et al., 2009; Yeh et al., 2013). From the above statement, it cleared that nutritional support is a crucial aspect of multi-modal cancer care, by improving the overall health status by suppressing various adverse events as well as enhance treatment regimen for a speedy recovery. Hence, the present multi-centered, randomized clinical trial was framed to evaluate the efficacy of ready to use balanced nutritional formula-PCNF (rich in ω-3 FA, fibers, MTC, BCAA, and micro-nutrients), in various cancer patient by checking calorie intake and overall health status through assessing various anthropometric and biochemical parameters especially total proteins, pre-albumin, and transferrin.

ELIGIBILITY:
Inclusion Criteria:

* only hospitalized cancer patients with risk of malnutrition and underweight (confirmed with BMI, protein, and pre-albumin level) and must be under NG tube feeding.

Exclusion Criteria:

* avoiding cancer patients under critical conditions, with cardiac, renal, and hepatic disorders. Also, heavy smokers, chronic or chain smokers, and pregnant/lactating women were not included.

Ages: 55 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Calorie intake | 12 weeks
  The mean value of calorie intake (energy) were significantly increased in PCNF supplemented subjects
Anthropometric parameters | 12 weeks
  BMI were markedly improved in PCNF intook subjects
Protein nutritional assessment index or nutritional status | 12 weeks
  Protein nutritional assessment index (total protein, pre-albumin , and transferrin) were significantly improved

SECONDARY OUTCOMES:
Glycemic indices | 12 weeks
  No significant changes in any of the glycemic indices or lipid profile PCNF groups

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Kun Wang, Ph.D, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
No, it's confidential